

## NCT04656990

SKIPping With PAX: An Integrated Gross Motor and Social-Emotional Skill Intervention

Approval date: 7/30/2019

Consent form



## Dear Parents:

I am an Associate Professor at the University of South Carolina. My expertise is teaching basic movements to keep children physically active throughout their life through an intervention program called Successful Kinesthetic Instruction for Preschoolers (SKIP). This year the University of South Carolina has developed a school-wide partnership with the Lexington 4 Early Childhood Center (LECC) to provide children the SKIP program at school.

By allowing your child to participate, we will test their current motor skills by asking them to perform fun skills like striking, kicking and catching (Test of Gross Motor Development Third Edition). Afterwards, we will provide SKIP to your child at LECC during the school day. At the end of the school year, we will then test your child again to see if their motor skills have improved. In testing your child, we will film them to assess their movement; however, each child will be assigned a number and will never be identified by name. All testing results will only be seen by myself, the school district, and the research team at the University of South Carolina. You may request your child's scores on each test and the video of your child if you would like them.

The SKIP program and study is important for children to develop movement skills throughout their life. This is the first year of a multiple year program at the Lexington 4 Early Childhood Center in sponsorship with the University of South Carolina Department of Physical Education funded by the National Institutes for Health. Through this program, we can provide children and families with movement education and physical activity twice weekly throughout the school year. Data obtained from this program will be used as evidence for applying for future grant funding for the Lexington 4 Early Childhood Center. We would love for your child to participate in this program. By returning this form, you consent for your child to participate.

| Thank you | | |
|-----------------------------|----------------------------|---------------|
| I GIVE PERMISSION FOR MY CH | HILD TO PARTICIPATE IN THE | SKIP PROGRAM. |
| Child' Name | Child's Teacher | |
| Your Name | Your Signature | Date |